CLINICAL TRIAL: NCT07034703
Title: Prospective Cohort of Patients Treated Using Neoadjuvant Modified FOLFIRINOX 6 Cycles for Potentially Resectable Pancreatic Duct Adenocarcinoma, Candidate for Participation in the PANACHE02 Clinical Trial PANACHE02-SC
Brief Title: Prospective Cohort of Patients Treated Using Neoadjuvant Modified FOLFIRINOX 6 Cycles for Potentially Resectable Pancreatic Duct Adenocarcinoma, Candidate for Participation in the PANACHE02 Clinical Trial
Acronym: PANACHE02-SC
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Rouen (Other)
Collaborators: Federation of Research in Surgery (FRENCH) (Other)
Responsible Party: Sponsor
Other Study IDs: 2022/0280/OB
Record Dates: First submitted 2025-05-30; First posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Resectable Pancreatic Duct Adenocarcinoma
Keywords: FOLFIRINOX

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- mFOLFIRINOX: patients treated using Neoadjuvant modified FOLFIRINOX 6 cycles for potentially resectable pancreatic duct adenocarcinoma,

SUMMARY:
The aim of our study is to build up biological, radiological and tissue collections so as to identify, at the time of diagnosis of pancreatic adenocarcinoma, multifactorial factors and/or biomarkers (tissue, plasma, radiomic) predictive of the success of the complete therapeutic sequence.

So we can distinguish 3 biological collections here :

* Collection for ctDNA assay on STRECK tubes
* Collection on PAXgene tubes
* Tissus collection

Considering the biology collection for ctDNA assay : blood samples will be taken on specific tubes before the start of neoadjuvant chemotherapy (C1), Before C2 and after C4 of neoadjuvant chemotherapy. For ctDN assay, 2x 10ml STRECK tubes will be taken at each point for each patient.

At the end of the study, aliquots will be sent to INSERM unit U1245 to be analyzed

Considering the biology collection on PAXgene tubes : 2,5 ml blood samples will be taken in PAXgene blood RNA tube before C1 for each patient

Considering tissue collection: pre-chemotherapy biopsies and surgical specimens will be preserved after resection. Tissue sample will be collected and preserved in the tumor bank of Rouen university hospital,

By collecting data for all screened patients (complete sequence in PANACHE02, NT failure (progression), randomization failure after surgery) at diagnosis (clinicobiological data, pre-NT biopsies, blood samples and imaging data) we first aim to refine patient selection for NT benefit with a multivariable signature approach and to identify biomarkers (blood, imaging) monitoring during the neoadjuvant phase that could be predictive of early detection for NT treatment failure.

We therefore believe that the constitution of such cohort is critical to address numerous unmet needs.

ELIGIBILITY:
Inclusion Criteria:

* Pancreatic adenocarcinoma, confirmed by a histocytological analysis
* Potentially resectable pancreatic adenocarcinoma (according to the NCCN classification; Version 2.2017). Resecability is evaluated on arterial-phase and portal-phase IV contrast-enhanced multislice CT scan of the pancreas (slice thickness: 2.5 mm), as evaluated in a multidisciplinary staff meeting including at least one radiologist and one expert surgeon.
* No previous chemotherapy
* Age 18 or over
* PS Grade 0 or 1
* Absolute neutrophil count > 1,500 mm3 platelet count > 100,000 mm3 creatinine clearance (according MDRD equation) > 50 ml/min, haemoglobin level > 10 g/dl (transfusions are authorized)
* Women of child-bearing age not having undergone a hysterectomy or tubal ligation - requirement for a pregnancy test (abnormal serum or urine beta-HCG level) before inclusion.
* Provision of informed, written consent

Exclusion Criteria:

* Pancreatic adenocarcinoma defined as locally advanced non-resectable or metastatic.
* Dihydropyrimidine dehydrogenase complete deficiency (uracilemia ≥ 150 ng/ml)
* Surgical or anaesthesiological contra-indications:

  * non-controlled congestive heart failure - non-treated angina - recent myocardial infarction (in the previous year) - non-controlled AHT (SBP >160 mm or DBP > 100 mm, despite optimal drug treatment), long QT
  * major non-controlled infection
  * severe liver failure
* Any medical, psychological or social situation that (in the investigator's opinion) could limit (i) the patient's compliance with the protocol or (ii) the ability to obtain or interpret data
* Pregnant or breastfeeding women and women of child-bearing age not using effective means of contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The PANACHE02 screening cohort study is a prospective national multicenter cohort study including patients with resectable pancreatic duct adenocarcinoma treated with neoadjuvant FOLFIRINOX.
  Of note, patients included in the PANACHE02 screening cohort study will be candidate for participation in the PANACHE02 phase II/III clinical trial to investigate risk-adapted adjuvant chemotherapy guided by the tumor stage
Sampling Method: Non-Probability Sample
Enrollment: 820 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2030-09 (Estimated); Study Completion 2032-01 (Estimated)

PRIMARY OUTCOMES:
factors and/or multifactorial biomarkers signature predictive of success of the complete therapeutic sequence | from enrollment to the first cycle of adjuvant treatment up to 2 months
  In relation with the primary objective the primary endpoint of the PANACHE02 screening cohort study is the success for the complete therapeutic sequence defined by the administration of at least 4 cycles of neoadjuvant modified FOLFIRINOX following by pancreatic tumor resection and at least one cycle of adjuvant treatment.
  A patient evaluable for the primary endpoint is a patient for whom we the success or the failure of the complete therapeutic sequence.
  A patient in success for the complete therapeutic sequence is a patient with an administration of at least 4 cycles of neoadjuvant modified FOLFIRINOX following by pancreatic tumor resection and at least one cycle of adjuvant treatment.
  A patient in failure for the complete therapeutic sequence is a patient with an administration of less than 4 cycles of neoadjuvant modified FOLFIRINOX and/or no resection and/or no adjuvant treatment administration.

SECONDARY OUTCOMES:
Overall Survival (OS) in the overall population and according to the complete therapeutic sequence status | through study completion, an average of 76 months
  Overall survival; OS will be calculated from the date of diagnosis to the date of death from any cause. Alive patients will be censored at the last date known to be alive, either during study treatment period or during follow-up period.
prognostic value of ctDNA at diagnosis for OS | through study completion, an average of 76 months
  extraction of ctDNA, then quantification by fluorimetry before being analyzed by digital PCR (dPCR)
prognostic value of ctDNA at diagnosis for event free survival, | through study completion, an average of 76 months
  Event-free survival (EFS) was used to evaluate the time to failure since diagnosis. A failure is defined as progression before surgery, unresectable or metastatic disease at surgical exploration and recurrence or death whatever occurred first after surgery. Alive patients with no failure will be censored at the last date known to be alive with no failure events, either during study treatment period or during follow-up period.
tissue, serum and imaging libraries (Biological database development) | through study completion, an average of 76 months
  Assess several methods to quantify tumor response and its prognostic value. If pertinent and reproducible, the best method may better select the patients most likely to beneficiate from a chemotherapy switch than the pTNM stage. Different approaches will be compared to refine the identification of good/bad responders.
factors associated with early recurrence for patients resected (< 12 months after surgical resection). | from surgical resection to the end of follow-up period at 28 months
  For patients resected, Disease Free Survival (DFS), is defined as the time from complete surgical resection to first documented event (cancer relapse, second malignancy, or death, whichever occurred first), or until last contact if no event occurs. Patients lost to follow-up were censored at last follow-up visit.
the rate of patients with access to adjuvant treatment | from enrollment to the adjuvant treatment period, an average of 5 months
  Rate of patients with access to adjuvant treatment
factors at diagnosis associated with the access to adjuvant treatment | from enrollment to the adjuvant treatment period at 5 months
safety and tolerance of the neoadjuvant chemotherapy | from enrollment to 90 days post operatively
  Safety and will be measured by the incidence and grade of AEs, SAEs, according to NCI-CTCAE v 5.0
overall morbidity of the neoadjuvant chemotherapy | from enrollment to 90 days post operatively
  Overall morbidity evaluated with DINDO-CLAVIEN at 30 days and 90 days post operatively The Clavien Dindo classification scale consists of several grades ranging from a postoperative event not requiring medical treatment Grade I to death Grade V (Grade I, II, IIIa, IIIb, IVa, IVb and V)
surgical morbidity and mortality rates | from enrollment to 90 days post operatively
  Surgical morbidity and mortality rates are evaluated with DINDO-CLAVIEN at 30 days and 90 days post operatively The Clavien Dindo classification scale consists of several grades ranging from a postoperative event not requiring medical treatment Grade I to death Grade V (Grade I, II, IIIa, IIIb, IVa, IVb and V)
value of the tumour response | from enrollment to the end of follow-up period at 28 months
  size, T stage; resection margins, criterion R; lymph node invasion, N stage
Number of patients with complete neoadjuvant sequence | from enrollment to the end of follow-up period at 28 months
  complete neoadjuvant sequence correspond to mFOLFIRINOX Cycles + curative surgery
evolution of health-related quality of life | from enrollment to the end of follow-up period at 28 months
  (EORTC QLQ-C30 and QLQ-PAN26 questionnaires)

CONTACTS AND LOCATIONS:
Overall Officials: Pr SCHWARZ, Principal Investigator — University Rouen Hospital
Locations (1):
- CHU de Rouen, Rouen, France, France

IPD SHARING:
Plan to Share IPD: Undecided